CLINICAL TRIAL: NCT03069209
Title: Transplantation of Specific Populations of Bone Marrow-Derived Stem Cells and Mesenchymal Stem Cells for the Treatment of Premature Ovarian Failure.
Brief Title: Autologous Bone Marrow-Derived Stem Cell Transplantation in Patients With Premature Ovarian Failure (POF)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stem Cells Arabia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-POF1
Record Dates: First submitted 2017-02-25; First posted 2017-03-03 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cells (Experimental): Intervention: Intraovarian transplantation of autologous purified bone marrow-derived stem cells and mesenchymal stem cells.
  Interventions: Biological: Stem Cells

INTERVENTIONS:
Biological: Stem Cells — Intraovarian transplantation of autologous purified bone marrow-derived stem cells and mesenchymal stem cells.

SUMMARY:
This is an open label, single arm, single center investigation to assess the safety and efficacy of purified adult autologous bone marrow derived specific populations of stem cells and mesenchymal stem cells injected into the ovaries (intraovarian injection), through a 12 week follow-up period. The investigators' chosen model of study is based on increasing the efficiency of the approach by choosing an autologous model which preserves the genetic composition of an individual that is vital in infertility conditions. Additionally the approach involves transplanting a combination of specific purified stem cell types which all aid in ovarian function recovery.

DETAILED DESCRIPTION:
Premature ovarian failure (POF) is characterized as hypergonadotropic ovarian failure mostly prevalent before age 40. It is astonishingly frequent and affects around 1% of women below the age of 40. The clinical findings include amenorrhea and abnormally high levels of luteinizing (LH) and follicle stimulating hormone (FSH). The etiology of POF is unidentified in the majority of cases. It can occur due to a combination of genetics, immunological diseases, and environmental factors. POF is characterized by lack of secondary follicles, arrested folliculogenesis, decreased estrogen levels, and female infertility.

Currently, no available therapeutic intervention has been verified effective in retrieving fertility in patients with POF. Several trials at ovarian stimulation are typically ineffective. Consequently, the diagnosis of POF can cause great physical and emotional distress among patients. Hence, there is serious need to develop innovative treatment plans for POF.

The latest research shows that reduced ovarian reserve is caused by aging of the niche rather than a defect in germ cell lines. Current scientific evidence suggests that bone marrow-derived mesenchymal stem cells (BMSCs) could repair injured tissues and holds great promise in treating many diseases including male and female infertility.

The uniqueness of this study is demonstrated in the transplantation of purified specific populations of autologous bone marrow derived stem cells and mesenchymal stem cells (BMSCs) into patients with POF without in vitro expansion or culture, with minimal manipulation. Stem cells are withdrawn and transplanted back into the patient on the same day of the procedure, thus presenting the highest safety and efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age : 20-39
* FSH>20

Exclusion Criteria:

* Thyroid dysfunction
* Immunological Conditions
* Past history of malignancy/cemotherapy/radiotherapy
* Infectious diseases: HIV+, hepatitis B+, C+
* Abnormal karyotype
* Previous surgical management of ovarian pathology
* Severe endometriosis

Ages: 19 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-06 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Return of menstrual cycle | 6 months
  Return of menses in a woman with previous ameneorrhea for at least 6 months before recruitment.

SECONDARY OUTCOMES:
Pregnancy | 12 months
  Occurrence of pregnancy during the 12 months follow-up period
FSH levels | 12 months
  Normalization of FSH levels
Follicular function | 12 months
  development of ovarian follicles to a size at least 18 mm in diameter
Endometrium thickness | 12 months
  Increase in endometrial thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Stem Cells Arabia, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided